CLINICAL TRIAL: NCT02841059
Title: The Association of Total Hysterectomy and Disorders of Female Pelvic Floor or Sexual Function: a Survey on Pelvic Floor Function and Sexual Life for Women After Different Type of Hysterectomy
Brief Title: The Pelvic Floor Function and Sexual Life of the Women After Different Type of Hysterectomy
Acronym: HYS-PF-QOL
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: HYS-SEX-QOL-POP
Record Dates: First submitted 2016-06-20; First posted 2016-07-21 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2016-07

CONDITIONS: Quality of Life; Urinary Incontinence; Pelvic Organ Prolapse
Keywords: quality of life; urinary incontinence; POP
MeSH Terms: conditions — Urinary Incontinence; Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Laparoscopic subtotal hysterectomy: women with benign gynecology disease and decided to receive laparoscopic subtotal hysterectomy (LSH) after discussion with her surgeon.
  Interventions: Procedure: LSH
- Laparoscopic CLSH: women with benign gynecology disease and decided to receive laparoscopic cervical ligament sparing hysterectomy (CLSH) after discussion with her surgeon.
  Interventions: Procedure: CLSH
- Laparoscopic AVH: women with benign gynecology disease and decided to receive laparoscopic assisted vaginal hysterectomy (LAVH) after discussion with her surgeon.
  Interventions: Procedure: LAVH

INTERVENTIONS:
Procedure: LSH — laparoscopic subtotal hysterectomy: LSH
  Other Names: laparoscopic subtotal hysterectomy: LSH
  Groups: Laparoscopic subtotal hysterectomy
Procedure: CLSH — laparoscopic cervical ligament sparing hysterectomy: CLSH
  Groups: Laparoscopic CLSH
Procedure: LAVH — laparoscopic assisted vaginal hysterectomy: LAVH
  Groups: Laparoscopic AVH

SUMMARY:
In this prospective, comparative non-randomized multiple teaching hospitals study, the investigators try to determine the relationship of total hysterectomy and Taiwanese female pelvic floor and sexual function from the view of epidemiology and clinical survey. This is an important issue that related to female autonomy, health care resources and even national health policy. The study results will help to understand whether there is unnecessary part in the current hysterectomy procedures and its potential health hazard.

DETAILED DESCRIPTION:
Women with benign gynecology disease and indicated for laparoscopic hysterectomy (laparoscopic subtotal hysterectomy: LSH, laparoscopic cervical ligament sparing hysterectomy: CLSH, laparoscopic assisted vaginal hysterectomy: LAVH) are invited and explained the details of the protocol by the surgeon. The types of hysterectomy are determined by the patient and the surgeon together after discussion. All participant have to sign the informed consent. The participant will be followed up for two years after surgery. Preoperative evaluation on uterine condition, pelvic floor, questionaires were recorded. The perioperative parameters including surgical time, blood loss, and postoperative parameters such as pain score, hospitalization etc were recorded. The postoperative evaluation on pelvic floor condition, questionaires etc were also recorded at different time points.

ELIGIBILITY:
Inclusion Criteria:

1. Patient who is indicated for hysterectomy due to benign gynecology disease. The participant's husband is also welcomed to join the survey of the sexual life questionnaire but this is not a necessary inclusion criteria.

Exclusion Criteria:

1. Suspect of or diagnosed as cancer patient
2. Age < 30 or > 50 years old
3. Menopausal woman or woman who is nulliparous
4. Patient with advanced pelvic floor prolapse (stage 2, 3, 4) including uterine prolapse, cystocele, enterocele, rectocele.
5. Patient with prominent urinary incontinence that affect social activity or suggested to have surgery by gynecologist or urologist.
6. Patient with severe medical diseases such as liver cirrhosis, heart failure, poor control diabetes mellitus etc.
7. Patient with severe pelvic inflammatory disease/tubo-ovarian abcess or pelvic endometriosis or history of severe pelvic adhesions.
8. Psychiatric patients
9. Patient with chronic lung disease such as bronchial asthma, bronchiectasis, chronic obstructive pulmonary disease and interstitial lung disease

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patient who is indicated for hysterectomy due to benign gynecology disease. The participant's husband is also welcomed to join the survey of the sexual life questionnaire but this is not a necessary inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Quality of life change | up to 12 months after hysterectomy
  Evaluate the change of quality of life by questionaire --WHOQOL-BREF Taiwan version, at preoperation,1,3,6 and 12 months after hysterectomy.

SECONDARY OUTCOMES:
Pelvic organ prolapse change | up to 24 months after hysterectomy
  evaluate by Pelvic Organ Prolapse Quantification System (POP-Q) at preoperation, 6,12 and 24 months after hysterectomy.
Urinary disorders change | preoperation and 3,6 and 12 months after hysterectomy
  evaluate by UDI-6 short form at preoperation,3,6 and 12 months after hysterectomy.
Sexual life change | preoperation and 3,6 and 12 months after hysterectomy
  short form of PISQ-9 approved by International Urogynecological Association, IUGA, at preoperation,3,6 and 12 months after hysterectomy.
Urinary incontinence status change | preoperation and 3,6 and 12 months after hysterectomy
  evaluate by IIQ-7 short form at preoperation,3,6 and 12 months after hysterectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Mun-Kun Hong, MD, Principal Investigator — Department of Obstetrics and Gynecology
Locations (4):
- Taiwan (4):
  - Dalin Tzu Chi Hospital, Chiayi City, Chiayi
  - Buddhist Tzu Chi General Hospital, Hualien City, Hualien
  - Mennonite Memorial Hospital, Hualien City, Hualien
  - Taipei Tzu Chi Hospital, Taipei, Taipei

IPD SHARING:
Plan to Share IPD: Undecided